CLINICAL TRIAL: NCT06288932
Title: An Outcome Study of Conventional Steroids Vs. Steroids Combined with Mycophenolate for the Management of Newly Diagnosed Immune Thrombocytopenia Purpura: a Cost Effective Measure in Developing Nations.
Brief Title: Outcome Study of Conventional Steroids Vs. Steroids Combined with Mycopehnolate in Newly Diagnosed Immune Thrombocytopenia Purpura.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBD/IRB-263/08-2023
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Immune Thrombocytopenia Purpura
Keywords: ITP; MMF
MeSH Terms: interventions — Mycophenolic Acid; Therapeutics

STUDY DESIGN:
Intervention Model Description: The study will comprise the newly diagnosed patients of Immune thrombocytopenia purpura aged 5-60 year. Patients will with a 1:1 ratio among the two group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mycophenolate Mofetil (MMF) Treatment (Experimental): Patients in this arm will receive Mycophenolate Mofetil (MMF) at a starting dose of 500mg twice daily along with Prednisolone.
  The pediatric dose of MMF will be calculated by 30mg/kg/day. Dose adjustment will be based on treatment response, with potential increases to 750mg twice daily or 1g twice daily.
  MMF will be administered for a specific duration, as determined by the study design.
  Interventions: Drug: Mycophenolate Mofetil (MMF) Treatment
- Standard Treatment Control (No Intervention): Patients in this arm will receive the standard treatment for ITP, which may include corticosteroids (prednisolone) commonly used for ITP management.The treatment regimen will be determined based on current standard guidelines and clinical practice.

INTERVENTIONS:
Drug: Mycophenolate Mofetil (MMF) Treatment — The first-line treatment of immune thrombocytopenia purpura with Mycophenolate Mofetil produced a significant response, a lowered likelihood of refractory ITP, a better outcome, and less financial burden.
  Other Names: Suprimun
  Arms: Mycophenolate Mofetil (MMF) Treatment

SUMMARY:
Immune thrombocytopenia Purpura (ITP) is an autoimmune condition delineated by humoral as well as cell mediated immune response against thrombocyte surface proteins GPIIb/IIIa receptors, affecting primary homeostasis leading to mucocutaneous bleeding.ITP is characterized by platelet count <100 x 109/L. The conventional line of treatment for newly diagnosed ITP is steroids but significant disadvantages have been associated with long term use and a high risk of relapse when reducing the dose. The addition of MMF to the first line treatment of ITP resulted in substantial response and a lower risk of refractory ITP with decreased financial burden and improved outcome.

DETAILED DESCRIPTION:
Immune Thrombocytopenia Purpura (ITP) is an acquired, immune-mediated disorder characterized by a severe decrease in peripheral thrombocyte count to less than 100 x 10⁹/L, leading to mucocutaneous bleeding. Our primary objective is to evaluate the efficacy of adding Mycophenolate Mofetil (MMF) alongside steroids in the first-line treatment of ITP, aiming for an enhanced therapeutic response, lower risk of refractory and chronic ITP, reduced financial burden, and improved overall outcomes.

The study aims to validate the efficacy and safety of MMF as a first-line treatment option for ITP while reducing the economic burden and risk of relapse associated with the condition

ELIGIBILITY:
Inclusion Requirements:

• Age: 5-60 years • Number of plates: <30x109

Exclusion Standards:

Pregnancy; lactation; hepatitis B and C; HIV-reactive individuals; and medication allergies

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Platelet count monitoring | assessed after 3 months and 6 months of treatment.
  Platelet count improvement, as assessed through regular monitoring and according to response criteria:
  The response criteria to the treatment described as follow:
  1. Complete response: Platelet count ≥ 100 x 10^ 9 /L
  2. Partial response: Platelet count 30≥ 100 x 10 ^9 /L
  3. No response: Platelet count 30 x 10^9 /

SECONDARY OUTCOMES:
Assessment of Health-Related Quality of Life questionnaire | 12 months
  Health-related quality of life questionnaire
Incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rukh-e- Zainub, Pharm-D,Mphil(enrolled), Principal Investigator — National Institute of Blood Diseases and Bone Marrow Transplantation; Shafaq Abdul Samad, MBBS,FCPS, Study Director — National Institute of Blood Diseases and Bone Marrow Transplantation; Dr.Iyad Naeem, Ph.D, Study Chair — KARACHI UNIVERSITY
Locations (1):
- National Institute of Blood Diseases and Bone Marrow Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No